CLINICAL TRIAL: NCT03785262
Title: Low Energy Surface Waves to Prevent Urinary Infections and Catheter Associated Symptoms Among Patients With Neurogenic Bladder Dysfunction
Brief Title: Low Energy Surface Waves for Neurogenic Bladder Patients With Indwelling Catheters
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to recruit
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 113221
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Neurogenic Bladder; Urinary Tract Infections
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham (Sham Comparator): Inactive uroshield device
  Interventions: Device: Sham Uroshield
- Active Uroshield (Experimental): Active uroshield device
  Interventions: Device: Uroshield

INTERVENTIONS:
Device: Uroshield — The Uroshield device sends out low-frequency ultrasound waves which run along the surface of the catheter.
  Arms: Active Uroshield
Device: Sham Uroshield — The sham Uroshield device is identical to the active machine, but it does not send out low-frequency ultrasound waves along the surface of the catheter.
  Arms: Sham

SUMMARY:
The Uroshield device is a commercially available device with two parts: a disposable actuator which attaches to the external portion of the catheter and a portable battery. The device sends out low-frequency ultrasound waves which run along the surfaces of the catheter. These acoustic waves prevent bacteria from adhering to the catheter and prevent the formation of biofilm. Our objective is to conduct a pilot study to determine if the UroShield device can reduce bacteriuria and catheter biofilm formation among neurogenic bladder patients with an indwelling catheter, as well as improve urinary quality of life and symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Spinal cord injury (>1 year), multiple sclerosis (>1 year), spina bifida, parkinsons (>1 year)
3. Indwelling catheter (urethral or suprapubic) for >3 months, and used as primary bladder management mechanism
4. >1 urinary tract infection in the last 12 months

Exclusion Criteria:

1. Intravesical botox in the last 6 months
2. Chronic antibiotic suppressive therapy
3. Active symptomatic UTI on day of randomization
4. Unable to understand written and spoken English
5. Prior/current utilization of the Uroshield device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Bacteriuria | 30 days
  Proportion with bacteriuria >10^5 cfu at day 30

SECONDARY OUTCOMES:
Neurogenic bladder symptom score (NBSS) | 30 days
  Validated symptom score that measures symptoms related to neurogenic bladder dysfunction and urinary quality of life. Total scale ranges from 0-74, and a lower number is considered a better outcome and represents lower symptom burden.
Patient subjective rating of amount of sediment/debris at the end of the 30 days | 30 days
Total bacterial cell counts | 30 days
Microbiome comparison of biofilms | 30 days
Scanning electron microscopy of biofilms | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- St Josephs Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan